CLINICAL TRIAL: NCT00111098
Title: A Multicenter, Single Arm Study Evaluating Once Monthly Darbepoetin Alfa Dosing In Subjects With Chronic Kidney Disease (CKD) Not Receiving Dialysis
Brief Title: Treatment for Subjects With Chronic Kidney Disease (CKD) Not Receiving Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20030153
Record Dates: First submitted 2005-05-17; First posted 2005-05-18 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2008-08

CONDITIONS: Kidney Disease
Keywords: Anemia; Chronic Kidney Disease (CKD)
MeSH Terms: conditions — Kidney Diseases; Anemia; Renal Insufficiency, Chronic | interventions — Darbepoetin alfa

ARMS (1):
- darbepoetin alfa (Experimental)
  Interventions: Drug: Darbepoetin Alfa

INTERVENTIONS:
Drug: Darbepoetin Alfa — QM administration for 28 weeks, adjusted as necessary to maintain Hb between 11.0 - 13.0 g/dL PFS concentrations: 20, 30, 40, 50, 60, 80, 100, 150, 200 and 300 mcg.

SUMMARY:
The proposed study is designed to test a novel dosing paradigm that would facilitate the treatment of anemia in CKD patients not on dialysis. Anemic patients who have achieved and maintained target hemoglobin (Hb) on every 2 weeks (Q2W) dosing of darbepoetin alfa will have the dosing interval extended to once monthly (QM) dosing. Extending the dosing interval for darbepoetin alfa to QM represents a major potential benefit to both patients with CKD and their caregivers.

ELIGIBILITY:
Inclusion Criteria: - Diagnosis of CKD and not expected to initiate dialysis for the duration of the study - Estimated glomerular filtration rate (eGFR): greater than or equal to 15 mL/min and less than or equal to 60 mL/min measured by the following modified Modification of Diet in Renal Disease (MDRD) equation 9, 10 : eGFR = 186 x [serum creatinine]-1.154 x [Age]-0.203 x [0.742 if subject is female] x [1.212 if subject is black] - Clinically stable, in the judgment of the investigator - Mean Hb greater than or equal to 11.0 g/dL to less than or equal to 13.0 g/dL (mean of 2 values drawn at least 3 days apart during the screening period) - Transferrin saturation (Tsat) greater than or equal to 15.0% - Serum vitamin B12 and folate levels above the lower limit of the normal range - Receiving stable Q2W subcutaneous (SC) doses of Aranesp® (darbepoetin alfa). A stable dose is defined as less than or equal to 25% change in dose over the 6-week period immediately prior to enrollment and with no missed doses in this period Exclusion Criteria: - Prior recipient or scheduled to receive a kidney transplant - Diastolic blood pressure (BP) greater than 110 mm Hg or systolic BP greater than 180 mm Hg during screening - Acute myocardial ischemia - Hospitalization for congestive heart failure or myocardial infarction within 12 weeks before enrollment - Parathyroid hormone level greater than 1500 pg/mL - Major surgery within 12 weeks before enrollment (excluding vascular access surgery) - Currently receiving antibiotic therapy for systemic infection - Known positive HIV antibody or positive hepatitis B surface antigen - Clinical evidence of current malignancy and/or receiving systemic chemotherapy/radiotherapy with the exception of basal cell or squamous cell carcinoma of the skin and cervical intraepithelial neoplasia - Red blood cell (RBC) transfusions within 8 weeks before enrollment - Androgen therapy within 8 weeks before enrollment - Systemic hematologic disease (e.g., sickle cell anemia, myelodysplastic syndromes, hematologic malignancy; myeloma; hemolytic anemia) - Any disorder that may impact (in the judgment of the investigator) the ability to give informed consent for participation in this study - Pregnant or breast-feeding women - All subjects must practice adequate contraception (in the judgment of the investigator) throughout this trial - Treatment with an investigational agent or device within 30 days before enrollment or scheduled to receive an investigational agent other than those specified by this protocol during the course of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2004-03; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects on QM darbepoetin alfa dosing maintained with a mean Hb greater than or equal to 11.0 g/dL during the evaluation phase | Entire Study

SECONDARY OUTCOMES:
To determine Hb values over the duration of the study | Entire Study
To determine darbepoetin alfa doses over the duration of the study | Entire Study
To assess the safety of darbepoetin alfa | Entire Study

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Agarwal AK, Silver MR, Reed JE, Dhingra RK, Liu W, Varma N, Stehman-Breen C. An open-label study of darbepoetin alfa administered once monthly for the maintenance of haemoglobin concentrations in patients with chronic kidney disease not receiving dialysis. J Intern Med. 2006 Dec;260(6):577-85. doi: 10.1111/j.1365-2796.2006.01723.x. PMID 17116009
- [Result] Silver MR, Agarwal A, Krause M, Lei L, Stehman-Breen C. Effect of darbepoetin alfa administered once monthly on maintaining hemoglobin levels in older patients with chronic kidney disease. Am J Geriatr Pharmacother. 2008 Jun;6(2):49-60. doi: 10.1016/j.amjopharm.2008.05.002. PMID 18675764
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/20030153.pdf